CLINICAL TRIAL: NCT06591728
Title: The Effects Of Dietary Protocatechuic Acid (PCA) On The Function And Structure Of Participants With Prosthetic Joint Infection (PJI) Before Revision Surgery, As Measured By Standard Biomarkers
Brief Title: PCA Loading Time Before Knee Prosthetic Joint Infection Revision
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Dean Reeves Clinic (Other)
Collaborators: Lanny Johnson, M.D. (Unknown); Leo Whiteside, M.D. (Unknown)
Responsible Party: Principal Investigator, Dr. Dean Reeves, Principal Investigator, Dr. Dean Reeves Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PCALoading-01
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Prosthesis-Related Infections
MeSH Terms: conditions — Prosthesis-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral PCA (Other)
  Interventions: Dietary Supplement: Oral PCA

INTERVENTIONS:
Dietary Supplement: Oral PCA — Administration of 1,000 mg BID of oral PCA in individuals with knee prosthetic joint infection prior to revision surgery

SUMMARY:
Proof of principle pilot study of the effect of dietary nutritional loading of protocatechunic acid (PCA) on the health and welfare of individuals with prosthetic joint infection (PJI), as measured by standard biomarkers

DETAILED DESCRIPTION:
Our purpose in the pre-surgery serial aspiration study is to determine the optimal PCA loading time duration for those with knee PJI with planned single or two stage revision.Our hypothesis, related to changes in structure and function as a result of PCA administration is that dietary nutritional loading of this nutraceutical PCA via the oral route will benefit the health and welfare of such a subject and alter the function and or structure of the human body having a PJI, as measured by improvemen in a pain biomarker, and one or more laboratory-based biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* More than 3 weeks after total knee arthroplasty
* One or more symptoms of injection, including redness, swelling, pain, increasing range of motion loss, fever, nausea, and loss of appetite.
* WBC count of aspiration >50,0000 cells per μL

Exclusion Criteria:

- Not willing to undergo blood draw and joint needle aspiration weekly up to 4 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Walking Pain 0-10 NRS | 0,1, 2, 3, and 4 weeks
  Walking pain change from time 0 to weekly follow-ups from 1-4
Change in CRP | 0,1, 2, 3, and 4 weeks
  Blood CRP change from time 0 to weekly follow-ups from 1-4
Change in ESR | 0,1, 2, 3, and 4 weeks
  Blood ESR change from time 0 to weekly follow-ups from 1-4
Change in WBC count in aspirate | 0,1, 2, 3, and 4 weeks
  Total WBC count change in periprosthetic aspirate
Bacterial colony count in aspirate | 0,1, 2, 3, and 4 weeks
  Colony count graded as 0 (No colonies), 1 (Few colonies), 2 (moderate growth) 3(heavy growth), and 4 (too numerous to count)

SECONDARY OUTCOMES:
CXCL9 | 0 and 3 months
  Change in Immunity Factor CXCL9 from 0 to 3 months
HbA1c | 0 and 3 months
  Change in HbA1c from 0 to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Reeves, Principal Investigator — K. Dean Reeves, M.D., P.A.